CLINICAL TRIAL: NCT07058376
Title: Clinical Research of Effectiveness and Safety of Herbal Medicine Strategy for Chronic Low Back Pain : A Prospective, Multicenter, Pragmatic Randomized Clinical Study
Brief Title: Clinical Research of Effectiveness and Safety of Herbal Medicine Strategy for Chronic Low Back Pain
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Jaseng Medical Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: JS-CT-2024-06
Record Dates: First submitted 2025-07-01; First posted 2025-07-10 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-11

CONDITIONS: Chronic Low-back Pain (cLBP)
Keywords: herbal medicine; chronic back pain

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Herbal Medicine Strategy Group (Experimental): Participants in this group will receive individualized herbal medicine prescriptions tailored to their clinical condition (symptoms, imaging, and response to treatment). Prescriptions, including type, dosage, and frequency, are determined by Korean medicine doctors based on clinical judgment. The herbal medicine will be taken orally for a total of 30 days, prescribed every 10 days over three clinic visits. All prescription details will be recorded in the CRF.
  Interventions: Procedure: Herbal Medicine Strategy
- Standard Korean Medicine Treatment Group (Active Comparator): Participants in this group will receive standard Korean medicine treatments for chronic low back pain, including acupuncture, electroacupuncture, cupping, infrared therapy, moxibustion, and physical therapy. Treatments are provided twice weekly for 5 weeks (maximum 10 sessions), with slight adjustments allowed depending on symptom severity. Treatment protocols are based on clinician judgment, and all interventions and points used are recorded.
  Interventions: Procedure: Standard Korean Medicine Treatment

INTERVENTIONS:
Procedure: Herbal Medicine Strategy — A pragmatic intervention involving tailored herbal prescriptions created by Korean medicine doctors. The specific composition, dose, and duration of herbal medicine vary per patient, and prescriptions are adjusted according to clinical response.
  Arms: Herbal Medicine Strategy Group
Procedure: Standard Korean Medicine Treatment — This includes the application of Korean medical procedures widely used for chronic low back pain:
  Acupuncture: Insertion of needles at 10-20 selected acupoints for 10-15 minutes.
  Electroacupuncture: Electrical stimulation at 3 Hz to 4 acupoints for 10-15 minutes.
  Infrared Therapy: Application of infrared rays from 30 cm for 10-15 minutes.
  Cupping: Wet or dry cupping at 2-4 points on the lower back.
  Moxibustion: Applied to two points near the painful area at 43±1°C for 10-15 minutes.
  Physical Therapy (ICT or TENS): Applied for 10-15 minutes focusing on the quadratus lumborum.
  Treatment frequency is 2 times/week for 5 weeks, but may be adjusted to 1-3 times/week depending on symptoms. Total number of sessions is limited to 10.
  Arms: Standard Korean Medicine Treatment Group

SUMMARY:
This study is a pragmatic multicenter randomized controlled trial evaluating the effectiveness and safety of herbal medicine strategy for chronic low back pain, using standard Korean medicine treatment as the control.

DETAILED DESCRIPTION:
0. Background Chronic low back pain (CLBP) is a common musculoskeletal disorder often managed in Korean medicine. This study aims to evaluate the effectiveness and safety of herbal medicine strategies for CLBP within a real-world clinical setting. It was initiated as part of a national research project to generate evidence for insurance coverage of herbal prescriptions.

1. Patient Recruitment and Screening Phase A total of 150 patients with CLBP lasting more than 3 months will be recruited across seven Korean medicine hospitals. Patients will be randomly assigned (1:1) to either the herbal medicine strategy group or the standard Korean medicine treatment group. Randomization will be prospective and pragmatic, with no pre-specified protocol for individual treatments.
2. Treatment and Evaluation Phase

   Experimental Group (Herbal Medicine Strategy): Participants receive individualized herbal prescriptions based on clinical judgment. Medication is prescribed every 10 days for a total of 30 days.

   Control Group (Standard KM Treatment): Participants receive acupuncture, electroacupuncture, cupping, moxibustion, infrared therapy, and physical therapy twice weekly for 5 weeks, with slight variations allowed based on symptom severity.

   Treatment details and frequencies will be recorded in CRFs and assessed during and after the intervention.
3. Follow-Up Phase Participants will be followed up after the treatment period to assess outcomes. Evaluation includes pain intensity, affected areas, quality of life, and treatment adherence.
4. Monitoring Although the study is investigator-initiated, third-party monitoring will be conducted in accordance with HRPP and Korean GCP guidelines to ensure protocol compliance and data integrity.

ELIGIBILITY:
Inclusion Criteria:

* Individuals experiencing low back pain for more than 3 months.
* Low back pain Numeric Rating Scale (NRS) score of 5 or higher.
* Aged 19 years or older and younger than 70 years.
* Individuals who voluntarily agree to participate in the clinical study and provide written informed consent.

Exclusion Criteria:

* Diagnosed with serious underlying conditions that may cause low back or radiating leg pain (e.g., spinal metastases, acute fractures, or vertebral dislocations).
* Presence of progressive neurological deficits or severe neurological symptoms.
* Pain primarily caused by non-spinal soft tissue conditions (e.g., tumors, fibromyalgia, rheumatoid arthritis, gout).
* Presence of other chronic diseases that may interfere with the treatment outcomes or their interpretation (e.g., stroke, myocardial infarction, kidney disease, diabetic neuropathy, dementia, epilepsy).
* Currently taking steroids, immunosuppressants, psychiatric medications, or other drugs that may affect study outcomes.
* Contraindications to acupuncture treatment or conditions making acupuncture unsafe: bleeding disorders, current anticoagulant therapy, or severe diabetes with high risk of infection.
* Contraindications to herbal medicine or conditions making its use unsafe: disorders or post-surgical conditions affecting drug absorption, severe hepatic or renal disease (AST, ALT, γ-GTP, or serum creatinine more than twice the upper normal limit at screening).
* Use of pain-altering medications such as Non-Steroidal Anti-Inflammatory Drugs (NSAIDs) or receipt of acupuncture treatment within 1 week prior to screening.
* Pregnant or breastfeeding women, or those planning pregnancy.
* Patients who underwent lumbar spine surgery within the last 3 months.
* Participation in another clinical trial within 1 month prior to screening, or plans to participate in another clinical trial during this study or within 6 months of screening.
* Difficulty in providing written informed consent.
* Any other condition judged by the investigator to make participation in the study inappropriate.

Ages: 19 Years to 69 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 150 (Estimated)
Dates: Start 2025-10-31 (Actual); Primary Completion 2026-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Low Back Pain Numeric Rating Scale (NRS) | Baseline(Week 0), Week 3, Week 5, Week 7, Week 12, Week 19, Week 26
  The primary outcome measure will be the change in the NRS score between Baseline and Week 7, which corresponds to the first follow-up visit after the end of treatment.
  The intensity of low back pain over the past week will be assessed using the NRS. In this scale, patients select a number from 0 to 10 that best represents their current level of discomfort (0 indicates no pain, and 10 indicates the worst pain imaginable).
Oswestry Disability Index (ODI) | Baseline(Week 0), Week 3, Week 5, Week 7, Week 12, Week 19, Week 26
  The primary outcome measure will be the change in the ODI score between Baseline and Week 7, which corresponds to the first follow-up visit after the end of treatment.
  The functional status of participants will be evaluated using the ODI questionnaire, which was developed to assess the degree of disability caused by low back pain. The ODI consists of 10 items, each rated on a 6-point scale from 0 to 5. The total score is summed and then divided by the maximum possible score (50 points for 10 items) to calculate a percentage. A higher percentage indicates a greater level of disability. A validated Korean version of the ODI will be used in this study.

SECONDARY OUTCOMES:
Radiating Leg Pain Numeric Rating Scale (NRS) | Baseline(Week 0), Week 3, Week 5, Week 7, Week 12, Week 19, Week 26
  The intensity of radiating leg pain over the past week will be assessed using the NRS. Participants will select a number from 0 to 10 that best represents their current level of discomfort (0 indicates no pain, and 10 indicates the most severe discomfort imaginable).
Low Back Pain and Radiating Leg Pain Visual Analogue Scale (VAS) | Baseline(Week 0), Week 7, Week 12, Week 19, Week 26
  The VAS consists of a 100 mm horizontal line where one end represents "no pain" and the other end represents "worst pain imaginable." Participants will mark a point on the line corresponding to the intensity of their low back pain and radiating leg pain during the past week.
Roland-Morris Disability Questionnaire-6 (RMDQ-6) | Baseline(Week 0), Week 7, Week 12, Week 19, Week 26
  The RMDQ-6 is a validated short-form version of the Roland-Morris Disability Questionnaire-24 (RMDQ-24) used to rapidly assess disability related to low back pain. It includes 6 items, and participants will respond based on their current condition. Higher scores indicate greater disability.
Patient Global Impression of Change (PGIC) | Week 7
  The PGIC is a 7-point scale used to subjectively assess the patient's overall impression of improvement. The scale includes the following categories:
  1. = Very much improved,
  2. = Much improved,
  3. = Minimally improved,
  4. = No change,
  5. = Minimally worse,
  6. = Much worse,
  7. = Very much worse.
EQ-5D-5L (EuroQol-5 Dimension, 5-Level) | Baseline(Week 0), Week 3, Week 7, Week 12, Week 19, Week 26
  The EQ-5D-5L is a widely used instrument for assessing health-related quality of life across five domains: mobility, self-care, usual activities, pain/discomfort, and anxiety/depression. Each item has five levels of response. Weighted values are applied to each level to compute an index score representing the individual's overall health state.
Health-related Quality of Life Instrument with 8 Items (HINT-8) | Baseline(Week 0), Week 3, Week 7, Week 12, Week 19, Week 26
  The HINT-8 is a Korean-specific instrument developed to measure health-related quality of life, covering physical, social, mental, and positive health dimensions. It includes 8 items: climbing stairs, pain, energy, work, depression, memory, sleep, and happiness.
  Participants will choose one of four response levels per item. For example, in the stair-climbing item:
  1. = No difficulty,
  2. = Some difficulty,
  3. = Severe difficulty,
  4. = Unable to climb stairs.
  For depression:
  1. = Not depressed at all,
  2. = Occasionally depressed,
  3. = Frequently depressed,
  4. = Always depressed.
Patient Health Questionnaire-15 (PHQ-15) | Baseline(Week 0), Week 7, Week 12, Week 19, Week 26
  The PHQ-15 is a validated Korean version of a 15-item questionnaire derived from the Patient Health Questionnaire (PHQ) used to assess general health status and somatic symptoms over the past 4 weeks. Each item is rated on a 3-point scale:
  0 = Not bothered at all,
  1. = Bothered a little,
  2. = Bothered a lot.
  The total score ranges from 0 to 30 and reflects symptom severity:
  0-4 = Minimal, 5-9 = Mild, 10-14 = Moderate, 15-30 = Severe. PHQ-15 is widely used to assess somatic symptom burden and is helpful in evaluating depression and somatoform disorders.
Credibility and Expectancy | Screening Visit
  Treatment expectation will be assessed using a 9-point Likert scale. At the screening visit, participants will be asked:
  "How much do you think traditional Korean medicine treatment will relieve your symptoms?"
  Response options range from:
  1 = Not at all, 5 = Somewhat, 9 = Very much.
Economic evaluation question | Baseline(Week 0), Week 3, Week 7, Week 12, Week 19, Week 26
  Cost data will be collected using a structured questionnaire designed to measure direct medical costs (e.g., medical services), non-medical costs (e.g., transportation, caregiver expenses), informal medical costs (e.g., health supplements, devices), and productivity losses. Productivity loss will be evaluated using the Work Productivity and Activity Impairment (WPAI) questionnaire, and economic costs will be estimated for cost-effectiveness analysis.
Drug Consumption | Baseline(Week 0), Week 3, Week 5, Week 7, Week 12, Week 19, Week 26
  Information on medications taken during the study period for current medical conditions will be collected at each visit, including drug name and dosage. Additionally, other treatments such as physical therapy or injections will be recorded by frequency.

OTHER OUTCOMES:
Adverse Events | Week 1, Week 2, Week 3, Week 4, Week 5, Week 7, Week 12, Week 19, Week 26
  Adverse events are defined as any undesirable and unintended signs (e.g., abnormal lab results), symptoms, or diseases occurring after study procedures, regardless of causality. Events will be collected through participant self-reports and investigator observation, and analyzed by frequency between groups.
  The relationship of each adverse event to the study treatment will be assessed using the WHO-UMC causality assessment scale:
  1. = Certain,
  2. = Probable/Likely,
  3. = Possible,
  4. = Unlikely,
  5. = Conditional/Unclassified,
  6. = Unassessable/Unclassifiable.
  Severity will also be categorized using Spilker's classification:
  Mild (1): No treatment needed; does not interfere with daily function.
  Moderate (2): Noticeable interference with daily function; may require treatment and recoverable.
  Severe (3): Requires intensive treatment; may result in sequelae.

CONTACTS AND LOCATIONS:
Overall Officials: In-Hyuk Ha, PhD, Principal Investigator — Jaseng Medical Foundation
Locations (1):
- Jaseng Hospital of Korean Medicine, Seoul, Gangnam-Gu, South Korea

IPD SHARING:
Plan to Share IPD: No